CLINICAL TRIAL: NCT03483142
Title: the Effect of Misoprostol on Intra-operative Blood Loss During Myomectomy Operation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ahmed nagy shaker ramadan (Other)
Responsible Party: Sponsor-Investigator, ahmed nagy shaker ramadan, resident of obstetric and gynecology, Ain Shams Maternity Hospital
Organization: Ain Shams Maternity Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Myomectomy
Record Dates: First submitted 2018-03-16; First posted 2018-03-30 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Myoma;Uterus; Blood Loss
MeSH Terms: conditions — Myofibroma; Hemorrhage | interventions — Misoprostol

STUDY DESIGN:
Intervention Model Description: Intervention
  All women will be randomly assigned to either:
  Group A ( study group ) ( 25 patient): who will receive placebo . two rectal placebo tablet of the same size and shape as the misoprostol.
  Group B (control group ) ( 25 patient): who will receive 400 microgram (tablet 200mcg X 2) misoprostol rectally one hour before operation
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- misoprostol group (Experimental): misoprostol group ( study group ) ( 25 patient): who will receive 400 microgram (tablet 200mcg X 2) misoprostol rectally one hour before operation
  Interventions: Drug: Misoprostol
- placebo group (Placebo Comparator): ( 25 patient): who will receive placebo . two rectal placebo tablet of the same size and shape as the misoprostol.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Misoprostol — ( 25 patient): who will receive 400 microgram (tablet 200mcg X 2) misoprostol rectally one hour before operation
  Other Names: misotac
  Arms: misoprostol group
Drug: Placebos — ( 25 patient): who will receive placebo . two rectal placebo tablet of the same size and shape as the misoprostol
  Arms: placebo group

SUMMARY:
assess the effect of using misoprostol in abdominal myomectomy operations on blood loss, duration of the operation and possible operative complications. Research question Does pre-operative misoprostol affect on intra-operative blood loss during and after myomectomy operation ?. Research hypothesis Pre-operative misoprostol may reduce intra-operative blood loss during and after myomectomy operation .

DETAILED DESCRIPTION:
. Type of Study : Prospective double blind randomized placebo controlled clinical trial.

* Study Setting : This study will be conducted in Ain Shams University Maternity hospital.
* Study Period : 6 months
* Study Population : Patients will be recruited in this study those attending gynecology ward at Ain Shams University Maternity hospital who are 25-50 years old with symptomatic uterine myoma

Methodology

All women will be subjected to:

History taking:

It includes name, age, occupation, marriage and special habits,last menstrual period, menstrual history, history of present illness ( symptoms related to myoma ), any medical disorders and any previous surgeries.

Examination

General examination:

It includes blood pressure, heart rate and body temperature, body mass index, head& neck examination Bilateral lower limb examination.

Abdominal examination:

It includes:

1. Inspection : pelvi-abdominal swelling
2. Palpation : smooth or irregular surface - mobility - consistency - size - tenderness
3. Auscultation : soufflé ( increased vascularity )
4. Percussion : dullness

Local examination:

Vaginal examnation will be done to detect uterine swelling with transmitted movement to the cervix . if movement not transmitted to cervix , it revealed extra-uterine swelling , also examination of adnexa Investigations Ultrasonography ( abdominal / vaginal ), (hysteroscopy , MRI , D&C if indicated ) Pre-operative investigation ( Complete blood picture, blood group , RH, hematocrite , Kidney Function Test , Liver Function Test , random Blood Sugar , urine analysis Intervention

All women will be randomly assigned to either:

Group A ( study group ) ( 25 patient): who will receive placebo . two rectal placebo tablet of the same size and shape as the misoprostol.

Group B (control group ) ( 25 patient): who will receive 400 microgram (tablet 200mcg X 2) misoprostol rectally one hour before operation

In all operations, the abdomen is entered by a Pfannenstiel incision. The operations are performed by the same team to avoid any bias related to surgical skills. The total volume of intra-operative blood loss is estimated by measuring the amount of blood accumulated in the suction container and the amount of blood on the surgical gauze by gauze weighting, the surgical gauzes are weighted before and after surgery using a scale accurate to 1 gram and the weight difference was calculated. The weight of 1 gram is taken as 1 ml blood.

Vital data during operation and the duration of the operation are recorded (time from opening of the peritoneum until its closure). The postoperative haemoglobin level is measured for each participant 24 h after the operation. Records are kept for any intra-operative or postoperative blood transfusion. Any postoperative adverse events, including any febrile episode (increase to or over 38.5°C in body temperature within 24 h following surgery) are documented. Also post operative vital data will be recorded

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal patients aged between 35 to 50 years old.
* Five or less symptomatic uterine myomas .
* Maximum diameter of the largest myoma is 6 cm .
* All myomas are subserous or intramural.
* Uterine size less than 24 weeks pregnancy

Exclusion Criteria:

* History of previous surgery.
* Allergy to Misoprostol.
* Hypertension.
* Cardiac and Pulmonary diseases.
* Patients who have bleeding disorders.
* Anemia (Hb < 10g %).
* Chronic endocrine or metabolic diseases such as Diabetes.
* Obesity (body mass index > 30 kg/m2).
* Cases that will require intraoperative conversion of myomectomy to hysterectomy.

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-07-30 (Estimated); Study Completion 2018-07-30 (Estimated)

PRIMARY OUTCOMES:
blood loss | time of operation
  reduce intra operative blood loss during myomectomy

CONTACTS AND LOCATIONS:
Overall Officials: sabry sayed, professor, Principal Investigator — Ain Shams Maternity Hospital
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Abbasia, Egypt